CLINICAL TRIAL: NCT05599581
Title: Tu'Washindi Randomized Control Trial (RCT): A Relationship-focused Intervention to Reduce Intimate Partner Violence (IPV) and Increase Pre-exposure Prophylaxis (PrEP) Uptake and Adherence Among Kenyan Adolescent Girls and Young Women (AGYW)
Brief Title: Tu'Washindi RCT: Adolescent Girls in Kenya Taking Control of Their Health
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Impact Research & Development Organization (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH12567
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: IPV; HIV; PrEP
Keywords: Adolescent Girls and Young Women (AGYW); Human Immunodeficiency Virus (HIV); Intimate Partner Violence (IPV); Kenya; Pre-exposure prophylaxis (PrEP)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Cluster-randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tu'Washindi intervention plus usual HIV prevention services (Experimental): Participants in the intervention wards will receive the Tu'Washindi intervention plus access to evidence-based HIV prevention services offered throughout the county. These include PrEP delivery through the Ministry of Health, which is accessible to all AGYW.
  Interventions: Behavioral: Tu'Washindi
- Standard of care HIV (Usual) prevention services only (No Intervention): Participants in the non-intervention (control) wards will have access to evidence-based standard of care HIV prevention services offered throughout the county. These include PrEP delivery through the Ministry of Health facilities, which is accessible to all AGYW.

INTERVENTIONS:
Behavioral: Tu'Washindi — Tu'Washindi consists of 3 primary components:
  1. PrEP Adherence Support Clubs: Eight 2-hour sessions that occur over the intervention period: twice per month for the first 2 months & once per month for the remaining 4 months. Sessions will use structured & unstructured activities designed to improve outcomes expectations, increase self-efficacy to use PrEP safely & consistently, increase peer support for PrEP use, provide access to community IPV resources & provide skills for healthy communication & PrEP disclosure with male partners.
  2. Community Male Sensitization conducted weekly over the first 3 months of the intervention period aimed to increase PrEP knowledge, reduce stigma, & promote healthy relationship communication.
  3. Buddy Days, which take place 3 months into the intervention period, designed to bring participants & their male partners together to learn about PrEP, discuss community attitudes & concerns regarding PrEP use, & promote HIV prevention & family well-being.
  Arms: Tu'Washindi intervention plus usual HIV prevention services

SUMMARY:
This study will test the effectiveness of a youth-designed multilevel intervention, Tu'Washindi, to increase PrEP use and reduce intimate partner violence (IPV) among Kenyan AGYW and to identify implementation challenges and strategies to facilitate future scale-up in programmatic settings to maximize public health impact.

Through a cluster randomized controlled trial (cRCT) design, twenty-two administrative wards in Siaya County, western Kenya will be randomized in a 1:1 ratio to receive either the 6-month Tu'Washindi intervention plus usual HIV prevention services or usual HIV prevention services alone. Approximately 72 AGYW will be enrolled from each ward (N= 1,584), with follow-up visits at months 3, 6, and 12 post-enrollment. A mixed methods process evaluation (not part of the clinical trial) will also be conducted using programmatic data, follow-up questionnaires from trial participants, approximately 500-1000 exit surveys with men, and approximately 100 qualitative interviews with AGYW participants, male partners, and intervention providers. These data will characterize fidelity and quality of intervention implementation, explore and test mechanisms of change, and capture contextual factors influencing intervention outcomes, with the goal of informing future refinement and implementation.

The population for this clinical trial study is AGYW ages 15-24 in Siaya County, Kenya.

DETAILED DESCRIPTION:
The Tu'Washindi intervention was developed to address factors at the individual, partnership, and community levels that influence AGYW's response to IPV and their PrEP use. These factors are addressed in a three-component intervention delivered over 6 months: a PrEP adherence support club for AGYW, PrEP education events for couples offered in the context of a health fair ("Buddy Days"), and community sensitization about PrEP targeted toward AGYW's partners.

The pilot cluster randomized controlled trial of Tu'Washindi intervention demonstrated feasibility, high acceptability, implementation with fidelity, and promising effects on PrEP and IPV outcomes. Importantly, AGYW perceived Tu'Washindi as effective in achieving its objectives: Nearly all participants agreed that Tu'Washindi improved communication and reduced conflict with their partner, and more than half reported that it helped them gain partner support for their PrEP use. Providers believed the intervention resonated with community values, integrated well within the scope of their ongoing responsibilities, and was feasibly integrated into existing HIV prevention programming. PrEP uptake and adherence were both twice as high in the intervention arm as in the control arm (p<0.05), and less frequent or severe IPV among intervention arm participants were observed.

This study will consist of a cRCT design with the primary objectives of testing the effectiveness of the Tu'Washindi intervention on PrEP uptake and adherence immediately at intervention endline and 6 months post-delivery (Aim 1) and secondary objectives of testing the effectiveness of the intervention on IPV (Aim 2). The study setting will be Siaya County located in the former Nyanza Province in western Kenya. Siaya County has the second highest HIV incidence in Kenya (2.5% per year) and the highest prevalence of IPV in Kenya (22% of women aged 15-49 have reported sexual violence and 56% have reported physical violence at least once since age 15).

Twenty-two administrative wards in Siaya will be randomized in a 1:1 ratio and enroll approximately 72 AGYW from each (total N= 1,584) to receive either the Tu'Washindi intervention plus usual HIV prevention services, or usual HIV prevention services alone. After informed consent and baseline data collection, the Tu'Washindi intervention will be implemented in each intervention cluster while the control cluster continues with usual HIV prevention services. Participants will be followed for 12 months, with data collection visits at intervention midline (Study Month 3), intervention endline (Study Month 6), and at 6 months post-intervention (Study Month 12).

A prospective process evaluation will be conducted to characterize intervention implementation, explore theorized mechanisms of change, and capture contextual factors influencing study outcomes (Aim 3). Although the cRCT will answer primary research questions about intervention effectiveness, the process evaluation will elucidate why and how the intervention was able to achieve these outcomes or suggest reasons for lack of any observed change. Additionally, it will provide important insight into how the intervention might be refined, adapted, and implemented in the future.

ELIGIBILITY:
Inclusion Criteria:

To join the study potential AGYW participants must be:

* Age 15-24 years
* Female
* Currently in a sexual relationship with a male partner for at least 1 month
* Susceptible to HIV per modified Determined, Resilient, Empowered, AIDS-free, Mentored and Safe (DREAMS) eligibility score
* (a) Taking PrEP or (b) interested in PrEP (i.e., thinks she would benefit from PrEP but is not currently taking it)
* Resident of applicable ward
* Willing and able to attend support clubs for over 6 months
* Willing and able to provide adequate contact information for retention
* Fluent in one of the study languages (English, Dholuo, or Kiswahili)
* (a) If aged 18 and above: Willing and able to provide informed consent; or (b) if non-mature minor aged 15-17: willing and able to provide assent and parent or guardian willing and able to provide parental consent; or (c) if mature minor aged 15-17: willing and able to provide informed consent or to provide assent and parent or guardian consent, per participant choice.

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Females
Enrollment: 1562 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Effective PrEP use (biomarker assessment) | 6-month follow-up
  Percent of all study participants with biomarker tenofovir-diphosphate levels indicating consistent PrEP use (≥4 doses per week) for the past 2 months measured as concentrations in dried blood spots. Represents a composite outcome of PrEP initiation, persistence, and high execution to capture these steps in the HIV prevention continuum.
Effective PrEP use (biomarker assessment) | 12-month follow-up
  Percent of all study participants with biomarker tenofovir-diphosphate levels indicating consistent PrEP use (≥4 doses per week) for the past 2 months measured as concentrations in dried blood spots. Represents a composite outcome of PrEP initiation, persistence, and high execution to capture these steps in the HIV prevention continuum.

SECONDARY OUTCOMES:
IPV prevalence | 3-month follow-up
  Percent of participants reporting IPV since the last study visit, measured with the World Health Organization (WHO) VAWI and classified by the Tackling the Structural Drivers of HIV (STRIVE) Consortium definition: any act of severe physical or sexual violence, or >=2 acts of moderate physical violence.
IPV prevalence | 6-month follow-up
  Percent of participants reporting IPV since the last study visit, measured with the World Health Organization (WHO) VAWI and classified by the Tackling the Structural Drivers of HIV (STRIVE) Consortium definition: any act of severe physical or sexual violence, or >=2 acts of moderate physical violence.
IPV prevalence | 12-month follow-up
  Percent of participants reporting IPV since the last study visit, measured with the World Health Organization (WHO) VAWI and classified by the Tackling the Structural Drivers of HIV (STRIVE) Consortium definition: any act of severe physical or sexual violence, or >=2 acts of moderate physical violence.
IPV severity | 3-month follow-up
  Percent of participants reporting any sexual or severe physical IPV since the last study visit, measured with WHO VAWI.
IPV severity | 6-month follow-up
  Percent of participants reporting any sexual or severe physical IPV since the last study visit, measured with WHO VAWI.
IPV severity | 12-month follow-up
  Percent of participants reporting any sexual or severe physical IPV since the last study visit, measured with WHO VAWI.
IPV intensity | 3-month follow-up
  Self-report continuous score calculated from the number of specific violent acts reported and the reported frequency of each act (0=never; 1=once; 2=a few times; 3=often) since the last study visit, measured with WHO VAWI.
IPV intensity | 6-month follow-up
  Self-report continuous score calculated from the number of specific violent acts reported and the reported frequency of each act (0=never; 1=once; 2=a few times; 3=often) since the last study visit, measured with WHO VAWI.
IPV intensity | 12-month follow-up
  Self-report continuous score calculated from the number of specific violent acts reported and the reported frequency of each act (0=never; 1=once; 2=a few times; 3=often) since the last study visit, measured with WHO VAWI.

CONTACTS AND LOCATIONS:
Locations (2):
- Kenya (2):
  - Impact Research and Development Organization (IRDO), Kisumu
  - RTI International Africa Regional Office, Nairobi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roberts ST, Minnis AM, Napierala S, Montgomery ET, Digolo L, Cottrell ML, Browne EN, Ndirangu J, Boke J, Agot K. Evaluation of the Tu'Washindi Na PrEP Intervention to Reduce Gender-Based Violence and Increase Preexposure Prophylaxis Uptake and Adherence Among Kenyan Adolescent Girls and Young Women: Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2025 Apr 1;14:e55931. doi: 10.2196/55931. PMID 40168655